CLINICAL TRIAL: NCT01430065
Title: A Phase 1, Open Label, Single Sequence, Drug Interaction Study of the Pharmacokinetics of ASP015K and Tacrolimus After Separate and Concomitant Administration to Healthy Adult Volunteers
Brief Title: Pharmacokinetic Interaction Study to Assess the Effect of ASP015K on Tacrolimus in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 015K-CL-PK02
Record Dates: First submitted 2011-06-30; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Pharmacokinetics of ASP015K; Drug Interactions; Healthy Subjects
Keywords: transplant; ASP015K; tacrolimus; Prograf; healthy volunteers
MeSH Terms: interventions — peficitinib; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus and ASP015K (Experimental)
  Interventions: Drug: ASP015K; Drug: Tacrolimus

INTERVENTIONS:
Drug: ASP015K — oral
Drug: Tacrolimus — oral
  Other Names: Prograf; FK506

SUMMARY:
This study characterizes the pharmacokinetic effects of ASP015K on Tacrolimus in healthy volunteers.

DETAILED DESCRIPTION:
The subjects will be confined to the unit for 13 days and have a brief follow-up visit to obtain hematology blood samples. Numerous blood and urine samples will be taken to determine the pharmacokinetics of the drugs.

ELIGIBILITY:
Inclusion Criteria:

* If female, the subject is at least 2 years post menopausal or is surgically sterile per documentation provided by a third party medical professional and the subject is not pregnant as documented by a negative serum pregnancy test
* If male, the subject agrees to sexual abstinence and/or to use a highly effective method of birth control during the study period
* Subject is medically healthy, with no clinically significant medical history or abnormalities observed upon physical examination or 12-lead electrocardiogram (ECG)
* Subjects must weigh at least 45 kg and have a body mass index (BMI) of 18-32 kg/m2

Exclusion Criteria:

* Subject has a history of chronic diarrhea
* Subject has been vaccinated within the last 60 days prior to study drug administration
* The subject has a previous history of any clinically significant neurological, gastro-intestinal, renal, hepatic, pulmonary, metabolic, cardiovascular, psychiatric, endocrine, hematological disorder or disease
* Subject has a positive test for hepatitis C antibody, or positive for hepatitis B surface antigen (HBsAg)
* Subject has a history of the human immunodeficiency virus (HIV) antibody
* The subject has an absolute neutrophil count (ANC) < 2500 cells/mm3 Subject has had clinically significant illness within 1 month prior to study drug administration
* Subject has a recent history (within the last 6 months) of drug or alcohol abuse or a positive urine screen for alcohol or drugs of abuse/illegal drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic assessment of AUC through the analysis of blood and urine samples | Up to Day 13

SECONDARY OUTCOMES:
Pharmacokinetic assessment of maximum concentration (Cmax) through the analysis of blood and urine samples | Up to Day 13

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States